CLINICAL TRIAL: NCT04288180
Title: Maladaptive Avoidance and Fear Conditioning in Social Anxiety Disorder
Brief Title: Social Anxiety Virtual Reality Study
Acronym: SAVR
Status: Terminated | Type: Observational
Why Stopped: COVID-19 Pandemic
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Tali Manber Ball, PhD, Instructor, Stanford University
Other Study IDs: IRB-48367
Record Dates: First submitted 2020-02-25; First posted 2020-02-28 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Social Anxiety Disorder
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Social Anxiety Disorder: A group of adults with social anxiety disorder will be recruited for a psychological/behavioral research study.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There will be no intervention in this study. Adults with social anxiety disorder will complete research assessments related to fear and safety learning.

SUMMARY:
This project aims to validate a virtual reality paradigm that assesses maladaptive avoidance behavior in social anxiety disorder. It also aims to generate a significant scientific advance by testing the hypothesis that maladaptive avoidance maintains anxiety through disruptions in safety learning.

DETAILED DESCRIPTION:
Although occasional mild social anxiety is a common human experience, social anxiety disorder has a devastating impact on patients' lives, leaving them vulnerable to medical, psychiatric, and socioeconomic complications. A key feature of social anxiety disorder is avoidance of social and/or performance situations in which judgment and evaluation from others might occur. Reducing avoidance is therefore an important treatment goal.

Despite the importance of avoidance, however, it is very difficult to assess a patient's tendency to avoid. Many prior assessments of avoidance measure adaptive (i.e., helpful) avoidance, in which an individual learns to avoid a truly noxious stimulus. However, anxiety disorders are characterized by maladaptive avoidance, in which a relatively safe stimulus is avoided resulting in interference with the individual's goals. In this study, the first aim is to validate a virtual reality paradigm to measure maladaptive avoidance behavior in adults with social anxiety disorder. The second aim is to test whether maladaptive avoidance behavior relates to safety learning (measured by a fear extinction task).

ELIGIBILITY:
Inclusion Criteria:

* age 18+
* primary diagnosis of social anxiety disorder
* fluent spoken and written English
* able to provide informed consent

Exclusion Criteria:

* history of manic episode, hypomanic episode, or psychosis
* moderate or severe substance use disorder in the past 12 months
* current major depressive episode greater than moderate severity (PHQ-9 score >14)
* high risk for suicide (>8 on the MINI Suicidality section and/or clinician judgment that immediate medical attention is necessary)
* general medical condition or impediment to vision, hearing, or motor function likely to interfere with assessments
* benzodiazepine use in the past 2 weeks
* cannabis use for anxiety management in the past 2 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with primary social anxiety disorder, community sample
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Maladaptive Avoidance Behavior | Baseline
  Latency (in milliseconds) to enter the quadrant of the avoidance task containing the image from the fear learning task

SECONDARY OUTCOMES:
Maladaptive Avoidance Behavior (alternate measure) | Baseline
  Amount of time (in milliseconds) spent in the quadrant of the avoidance task containing the image from the fear learning task
Maladaptive Avoidance Behavior (2nd alternate measure) | Baseline
  Amount of time (in milliseconds) with center of gaze on the image from the fear learning task

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Undecided